CLINICAL TRIAL: NCT05448599
Title: A Study to Evaluate Pharmcokinetics, Pharmacodynamics , Efficacy and Safety of 6MW3211 Monotherapy and in Combination With Azacitidine(AZA) or AZA Plus Venetoclax(VEN) in Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: A Clinical Study of 6MW3211 Monotherapy or Combination Therapy for AML or MDS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6MW3211-2022-CP102
Record Dates: First submitted 2022-06-08; First posted 2022-07-07 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6MW3211 (Experimental): Phase I, 6MW3811 monotherapy in 2 dose levels of 30mg/kg or 45mg/kg; phase II, 6MW3811 will be given in combination with AZA( cohort1) and AZA plus VEN(cohort 2)
  Interventions: Drug: 6MW3211 injection with Intravenous Infusion

INTERVENTIONS:
Drug: 6MW3211 injection with Intravenous Infusion — phaseI: 6MW3211 will be administered in 30mg/kg and 45mg/kg intravenously once every 2 weeks; phaseII: 6MW3211 will be administered in 45mg/kg intravenously in both 2 cohorts.AZA will be administered in 75mg/m2 by subcoutaneous injection in cohort 1 as well as cohort 2 from Day1-Day7 every 28-day cycle. VEN will be administered orally with dose escalation to 400mg daily every cycle.
  Other Names: infusion

SUMMARY:
This study is aimed to evaluate the efficacy, safety, immunogenicity and pharmkinetics, pharmacodynamics of 6MW3211 as monotherapy and in combination with AZA or AZA plus VEN in patients with AML/MDS.

DETAILED DESCRIPTION:
This study is a phase I/II study to evaluate the pharmacokinetics, pharmacodynamics, efficacy and safety of 6MW3211 monotherapy or combined with AZA or AZA plus VEN in patients with AML and MDS. There will be 2 parts of this study. The phase Ib is about monotherapy of 6MW3211 and Phase II is designed to evaluate the safety and efficacy of 6MW3211 combined with AZA or AZA plus VEN in patients with relapse/refractory and newly diagnosed AML and MDS.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and sign the informed consent;
* 18≤age≤75，Men or women；
* AML patients (except acute promyelocytic leukemia) : subjects who meet the diagnostic criteria for relapsed/refractory AML according to the diagnostic criteria of 2021 Chinese Guidelines for the Diagnosis and Treatment of Relapsed and Refractory AML ； MDS patients: MDS patients were diagnosed as having moderate risk of recurrence/refractory (IPSS-R score >3.5) according to WHO diagnostic criteria in 2016
* ECOG:0-2;
* Survival expectation of at least 3 months;
* Adequate organs and hematopoietic functions; only applicable for phase II :
* Newly diagnosed AML with intolerance to standard induction chemotherapy who should meet one of following criterias: age ≥75 years; ECOG 2-3; chronic heart failure requiring treatment or EF≤50% or chronic stable angina pectoris; DLCO≤65% or FEV1≤65%;30ml/min≤CrCl<45ml/min；1.5 x ULN<total bilirubin≤3.0 x ULN
* Newly diagnosed intermediate- and high-risk (International Prognostic Scoring System IPSS-R) MDS

Exclusion criteria:

* Myeloid proliferative diseases (MPN), including primary myelofibrosis (PMF), polycythemia vera (PV), chronic myelogenous leukemia (CML), and primary thrombocytopenia (ET); Or have myelodysplastic myeloid proliferative tumors (MDS-MPN), including chronic monocytic leukemia (CMML), atypical chronic myelogenous leukemia (aCML), juvenile granulomatous single-cell leukemia (JMML), and acute promyelocytic leukemia (M3);
* Recurrence after allogeneic hematopoietic stem cell transplantation, or autologous hematopoietic stem cell transplantation within 1 year;
* Known infiltration of central nervous system leukemia；
* Active or uncontrolled autoimmune diseases；
* Has a history of other malignancies；
* Has known inherited or acquired hemorrhagic disorders；
* Pregnant or lactating women；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
CCR | 1 year
  Compound complete response rate
ORR | 1 year
  Objective Response Rate
phase II: safety | Up to 28 days post last dose
  to evaluate the percentage of participants with adverse events and serious adverse events of 6MW3211 combination therapy in AML and MDS

SECONDARY OUTCOMES:
AE | Up to 28 days post last dose
  All the adverse events
DoCR | 1 year
  Duration of complete response
RFS | 1 year
  Relapse-free survival
EFS | 1 year
  Event-free survival
OS | 1 year
  Overall survival
PK Parameter | 1 year
  The area under the curve (AUC)
Cmax | 1 year
  Maximum concentration
Tmax | 1 year
  Time at which maximum concentration
T1/2 | 1 year
  The half life

CONTACTS AND LOCATIONS:
Overall Officials: Hu Zhou, Ph.D, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No